CLINICAL TRIAL: NCT05458141
Title: DVx - SCHOOL: Digital Vaccine for Scalable Curricular Health Outcome Optimization and Learning
Brief Title: The Study Estimates the Longitudinal Impact of a Gamified Health Education App on Students' Health and Learning Outcomes
Acronym: DVx-SCHOOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Collaborators: University of Michigan (Other); Voluntary Health Services Hospital, Chennai, India (Unknown); Johns Hopkins Bloomberg School of Public Health (Other); FriendsLearn (Industry); University of Oxford (Other)
Responsible Party: Principal Investigator, Rema Padman, Trustees Professor Of Management Science And Healthcare Informatics, Carnegie Mellon University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: VHS/IEC/143/2022
Record Dates: First submitted 2022-07-07; First posted 2022-07-14 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-02

CONDITIONS: Infectious Disease; COVID-19; Physical Inactivity; Health Behavior; Nutrition, Healthy; Habit, Diet
Keywords: Digital Vaccine; Mobile Games; Physical Activity; Lifestyle Habit Formation; Infectious Diseases; Nutrition
MeSH Terms: conditions — Communicable Diseases; COVID-19; Sedentary Behavior; Health Behavior; Feeding Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Usual Education + Weekly Exposure to FYA-003 (Experimental): Students in grades assigned to Group 1 play FYA-003 in the classroom for 30 minutes every week for 12 weeks on a day at a time determined by the school & research team.
  Interventions: Behavioral: FYA-003
- Group 2: Usual Education + Weekly exposure to non-health related educational mobile games (No Intervention): Students in grades assigned to Group 2 play educational games unrelated to health in the classroom for 30 minutes every week for 12 weeks on a day at a time determined by the school & research team.

INTERVENTIONS:
Behavioral: FYA-003 — FYA-003: It is a gamified health education module for children aimed at promoting healthy nutrition, physical activity, health hygiene, and infectious diseases risk reduction within the clinically proven app fooya!
  Arms: Group 1: Usual Education + Weekly Exposure to FYA-003

SUMMARY:
The primary aim of this study is to assess and quantify the longitudinal impact of a mobile App-based module - FYA-003 - which is a gamified health education module for children promoting nutrition, physical activity, health hygiene, and infectious disease risk reduction within the clinically proven app fooya!, on the dietary and physical activity habits, hygiene practices, clinical outcome measures, and related knowledge of children and their caregivers. The app will be delivered in the classroom setting through school-based health education.

DETAILED DESCRIPTION:
A 2-arm cluster randomized controlled trial with pre-, during- and post-treatment measurements will be conducted in a school in Chennai (India) - Panchayat Union Middle School (PUMS), Katchipedu - to assess and quantify the longitudinal impact of a proposed Digital Vaccine candidate, called FYA-003®, on students' knowledge, behaviors and outcomes related to diet, physical activity and health hygiene. After following the protocol for recruitment and informed consent, the investigators will pair up grades in the school (site) in consecutive order, such as grades 1-2, 3-4, 5-6, and 7-8, and randomly assign one grade in the pair to Group 1 and the other to Group 2. These pairs are assumed to be close to each other in age, maturity levels, health related knowledge, and exposure to mobile apps, hence appropriate for pairing up for the study.

A team of research staff located in Chennai will coordinate the execution of the experiment. After following the protocol for participation by the school administrator and staff, and the protocol for student recruitment and informed consent, the investigators will adopt a cluster-randomized trial design, where treatment assignment will be done at the grade level. Actual food choice, clinical measurements, survey data, and food logs will be collected by the site PI with support from a research project coordinator during weekly visits to the school. Game play data will be collected automatically whenever the mobile device is connected to the internet and will be downloaded to a secure server after the school visits. The research team will coordinate the gameplay timing with the school officials.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-14
* Parents willing to participate (fill out parent surveys)

Exclusion Criteria:

* Children physically unable to use a device
* Children with special needs

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Health Knowledge Score - Baseline | Baseline
  Our primary outcome of interest is the health knowledge score, calculated based on students' survey responses to questions testing their knowledge on health hygiene, physical activity, and nutrition. This will be measured as a percentage. Higher percentages indicate a better outcome.
Health Knowledge Score - Week 4 | Week 4
  Our primary outcome of interest is the health knowledge score, calculated based on students' survey responses to questions testing their knowledge on health hygiene, physical activity, and nutrition. This will be measured as a percentage. Higher percentages indicate a better outcome.
Health Knowledge Score - Week 8 | Week 8
  Our primary outcome of interest is the health knowledge score, calculated based on students' survey responses to questions testing their knowledge on health hygiene, physical activity, and nutrition. This will be measured as a percentage. Higher percentages indicate a better outcome.
Health Knowledge Score - Week 12 | Week 12
  Our primary outcome of interest is the health knowledge score, calculated based on students' survey responses to questions testing their knowledge on health hygiene, physical activity, and nutrition. This will be measured as a percentage. Higher percentages indicate a better outcome.
Health Knowledge Score - Week 12 + 3mo | 3 months after Week 12
  Our primary outcome of interest is the health knowledge score, calculated based on students' survey responses to questions testing their knowledge on health hygiene, physical activity, and nutrition. This will be measured as a percentage. Higher percentages indicate a better outcome.
Health Knowledge Score - Week 12 + 6mo | 6 months after Week 12
  Our primary outcome of interest is the health knowledge score, calculated based on students' survey responses to questions testing their knowledge on health hygiene, physical activity, and nutrition. This will be measured as a percentage. Higher percentages indicate a better outcome.
Healthy Food Choice Score - Baseline | Baseline
  Observed "Good Food" choice indicator, as measured based on actual food choices by participants. This is a binary 0-1 value. 1 indicates a better outcome.
Healthy Food Choice Score - Week 4 | Week 4
  Observed "Good Food" choice indicator, as measured based on actual food choices by participants. This is a binary 0-1 value. 1 indicates a better outcome.
Healthy Food Choice Score - Week 8 | Week 8
  Observed "Good Food" choice indicator, as measured based on actual food choices by participants. This is a binary 0-1 value. 1 indicates a better outcome.
Healthy Food Choice Score - Week 12 | Week 12
  Observed "Good Food" choice indicator, as measured based on actual food choices by participants. This is a binary 0-1 value. 1 indicates a better outcome.
Healthy Food Choice Score - Week 12 + 3mo | 3 months after Week 12
  Observed "Good Food" choice indicator, as measured based on actual food choices by participants. This is a binary 0-1 value. 1 indicates a better outcome.
Healthy Food Choice Score - Week 12 + 6mo | 6 months after Week 12
  Observed "Good Food" choice indicator, as measured based on actual food choices by participants. This is a binary 0-1 value. 1 indicates a better outcome.

SECONDARY OUTCOMES:
Clinical biomarkers: BMI Baseline | Baseline
  Body Mass Index of participants
Clinical biomarkers: BMI Week 12 | Week 12
  Body Mass Index of participants
Clinical biomarkers: BMI Week 12 + 3mo | 3 months after Week 12
  Body Mass Index of participants
Clinical biomarkers: BMI Week 12 + 6mo | 6 months after Week 12
  Body Mass Index of participants
Clinical biomarkers: Average Temperature | Captured every week (Week 1 - Week 12)
  Average temperature of participants captured every weekly visit
Food Log Health Score - Baseline | Baseline
  Proportion of "Healthy" food items consumed in the weekly food logs recorded by the participants. Scale of 0 to 100. Higher score means better outcomes.
Food Log Health Score - Week 4 | Week 4
  Proportion of "Healthy" food items consumed in the weekly food logs recorded by the participants. Scale of 0 to 100. Higher score means better outcomes.
Food Log Health Score - Week 8 | Week 8
  Proportion of "Healthy" food items consumed in the weekly food logs recorded by the participants. Scale of 0 to 100. Higher score means better outcomes.
Food Log Health Score - Week 12 | Week 8, Week 12, 3 months after Week 12, 6 months after Week 12
  Proportion of "Healthy" food items consumed in the weekly food logs recorded by the participants. Scale of 0 to 100. Higher score means better outcomes.
Food Log Health Score - Week 12 + 3mo | 3 months after Week 12
  Proportion of "Healthy" food items consumed in the weekly food logs recorded by the participants. Scale of 0 to 100. Higher score means better outcomes.
Food Log Health Score - Week 12 + 6mo | 6 months after Week 12
  Proportion of "Healthy" food items consumed in the weekly food logs recorded by the participants. Scale of 0 to 100. Higher score means better outcomes.
Healthy Lifestyle Score - Baseline | Baseline
  Self-reported Weekly Healthy Lifestyle Score measured on the basis of participant survey responses to questions on physical activity, nutrition behavior, hygiene habits. Scale of 0 to 100. Higher score means better outcomes.
Healthy Lifestyle Score - Week 4 | Week 4
  Self-reported Weekly Healthy Lifestyle Score measured on the basis of participant survey responses to questions on physical activity, nutrition behavior, hygiene habits. Scale of 0 to 100. Higher score means better outcomes.
Healthy Lifestyle Score - Week 8 | Week 8
  Self-reported Weekly Healthy Lifestyle Score measured on the basis of participant survey responses to questions on physical activity, nutrition behavior, hygiene habits. Scale of 0 to 100. Higher score means better outcomes.
Healthy Lifestyle Score - Week 12 | Week 12
  Self-reported Weekly Healthy Lifestyle Score measured on the basis of participant survey responses to questions on physical activity, nutrition behavior, hygiene habits. Scale of 0 to 100. Higher score means better outcomes.
Healthy Lifestyle Score - Week 12 + 3mo | 3 months after Week 12
  Self-reported Weekly Healthy Lifestyle Score measured on the basis of participant survey responses to questions on physical activity, nutrition behavior, hygiene habits. Scale of 0 to 100. Higher score means better outcomes.
Healthy Lifestyle Score - Week 12 + 6mo | 6 months after Week 12
  Self-reported Weekly Healthy Lifestyle Score measured on the basis of participant survey responses to questions on physical activity, nutrition behavior, hygiene habits. Scale of 0 to 100. Higher score means better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Rema Padman, PhD, Principal Investigator — Carnegie Mellon University
Locations (1):
- Panchayat Union Middle School, Kanchipuram, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kato-Lin YC, Kumar UB, Sri Prakash B, Prakash B, Varadan V, Agnihotri S, Subramanyam N, Krishnatray P, Padman R. Impact of Pediatric Mobile Game Play on Healthy Eating Behavior: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Nov 18;8(11):e15717. doi: 10.2196/15717. PMID 33206054